CLINICAL TRIAL: NCT03219203
Title: Immunologic Response of Hepatitis B Single Dose Versus 3-dose Series in Previously Vaccinated HIV-infected Adults at Maharaj Nakorn Chiang Mai Hospital: A Randomized Controlled Trial
Brief Title: Immunologic Response of Hepatitis B Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4564
Record Dates: First submitted 2017-07-06; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis B
Keywords: HBV vaccination; immunity
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Single dose hepatitis B vaccine (Experimental): Single dose of hepatitis B vaccine group will receive a 20 µg recombinant HBV vaccine intramuscular at entry
  Interventions: Biological: Hepatitis B vaccine
- Arm B: 3-dose series of hepatitis B vaccine (Active Comparator): 3-dose series of hepatitis B vaccine group will receive a 20 µg recombinant HBV vaccine intramuscular at month 0, 1, and 6
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Hepatitis B vaccine — Hepatitis B vaccine (20 µg/ml) 1 ml intramuscular injection in single (at 0 month) or 3-dose series (at 0, 1, 6 months)

SUMMARY:
This study aims to evaluate the immunologic response to the two hepatitis B virus (HBV) vaccination booster strategies in previously vaccinated HIV-infected adults at Maharaj Nakorn Chiang Mai Hospital.

DETAILED DESCRIPTION:
This study intended to evaluate the immunologic response to the two hepatitis B virus (HBV) vaccination strategies in previously vaccinated HIV-infected adults at Maharaj Nakorn Chiang Mai Hospital.

As a part of HBV prevention program, HBV vaccine has been included in Thailand expanded program on immunization (EPI) since 1992. HBV vaccine has been shown to be safe, effective, and has a prolonged protective immunity to HBV infection. Despite the immunity from HBV vaccination could wane overtime, the previous data in general population revealed that HBV vaccine booster could raise the immune in very well. However, the data about booster effects for HBV vaccine among HIV-infected population who previously received a vaccination during their childhood is lagging. Based on previous data of vaccination response in HIV-infected population, the investigators estimate that the protective antibody will rise up to 60% with HBV vaccine one dose booster versus 90% with 3-dose series. Eighty participants, HIV-infected person who were born after HBV vaccine were born after HBV has been included in Thai EPI without evidence of HBV infection nor protective immunity, will be enrolled to this study (with estimation of 5% loss follow up rate). The participants will be randomized in 1:1. The immune response and vaccine safety will be evaluated at 1,7 and 12 months after the first dose HBV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Document of HIV infection
* Thai nationality
* Age ≥18 years old
* Born after 1 January 1992
* Has been taking antiretroviral drugs for HIV treatment
* CD4 ≥200 cell/mm3 and VL <50 copies/mL for at least 6 months before enrollment
* Negative for any HBV and HCV serological markers
* Willing to sign informed consent
* Able to follow up

Exclusion Criteria:

* Active opportunistic infection
* Pregnancy or breast feeding
* History of previous hepatitis B vaccine booster
* History of hypersensitivity to any component of vaccine
* Malignancy which received chemotherapy or radiation
* Immunocompromised condition such as solid-organ transplantation, chemotherapy in the last 6 months
* On Immunosuppressive treatment, immunomodulating treatment or general corticotherapy (equal or above 0.5 mg per kg per day )
* Renal failure (creatinine clearance <30 mL/min)
* Transaminitis in the past 3 months (≥ 5 UNL)
* Decompensated cirrhosis (child-Pugh class C)
* Unable or not willing to return for follow up

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Immunologic response to single dose versus 3-dose series of HBV vaccination in HIV-infected adults | 28 weeks after the first dose of HBV vaccination
  Immunologic response to single versus 3-dose series of HBV vaccination in HIV-infected adults, demonstrated by percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL ) at week 28

SECONDARY OUTCOMES:
Anamnestic response at week 4 | 4 weeks after the first dose of HBV vaccination
  Anamnestic response at week 4, demonstrated by percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL )
Percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL) at month 12 | 12 months after the first dose of HBV vaccination]
  Percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL) at month 12
Intensity and frequency of vaccine adverse event (AE) | 1 year
  Intensity and frequency of vaccine adverse event (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of medicine, Chiang Mai University, Muang, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No